CLINICAL TRIAL: NCT00956852
Title: Study on Systemic and Airway Cytokines and Oxidative Stress in Patients With Non-small Cell Lung Cancer (NSCLC) Undergoing Surgical Lung Resections
Brief Title: Study on Systemic and Airway Cytokines and Oxidative Stress in Lung Cancer Patients Undergoing Surgery
Status: Terminated | Type: Observational
Why Stopped: Poor subject recruitment
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Chung-Man HO, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 08-249
Record Dates: First submitted 2009-08-09; First posted 2009-08-11 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, buffy coat, red blood cell and exhaled breath condensate samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung cancer: Non-small cell lung cancer patients undergoing surgical lung resections

SUMMARY:
Lung cancer has remained as the top cancer killer in Hong Kong. Even for early resectable stage of lung cancer, only around 60-70% of patients can survive for 5 years after operation, mostly related to disease recurrence. Therefore there is urgent need for predictive biomarkers that can potentially help in monitoring patients for risk of disease recurrence after operation. Recent studies have suggested an important role of oxidative stress in the development of lung cancer and our preliminary data have suggested that some of the oxidative stress markers in blood could be predictive of response to systemic chemotherapy for lung cancer. Apart from potential biomarkers from blood, ongoing study has also been conducted to investigate the predictive role of biomarkers in exhaled breath condensate in lung cancer patients undergoing chemotherapy. Exhaled breath condensate can be collected simply with a disposable commercially available device that allows trapping of breath condensate via a cooling column during normal breathing for 20 minutes. Therefore this study aims at investigating the role of blood and exhaled breath condensate oxidative stress biomarkers before and after surgical lung resection for lung cancer in predicting subsequent clinical outcome, i.e., timing of disease recurrence. Recruited subjects will undergo interval sampling of blood and exhaled breath condensate, without any additional invasive interventions. The study subjects will be followed up for 5 years for subsequent disease recurrence.

DETAILED DESCRIPTION:
Lung cancer is the major cause of cancer deaths among both genders in Hong Kong. In 2005, primary lung cancer accounted for 33% and 25% of all cancer deaths in men and women respectively. On average, there are around 4,000 new cases of lung cancer each year. Non-small cell lung cancer (NSCLC) accounts for about 80% of all primary lung cancers. About 60% of cases present as advanced stages IIIB and IV disease. The currently available treatment modalities include surgery, radiotherapy and systemic chemotherapy. However, the overall prognosis remains dismal with 5-year survival rate less than 15%. Among those with early stage lung cancer, the 5-year survival rate is still suboptimal at around 60-70%. Therefore, there has been immense interest in the development of novel biomarkers to delineate the high risk group for subsequent tumour recurrence after curative lung resections. It has long been found that cellular prooxidant states promote cells to neoplastic growth, in part due to DNA damage caused by reactive oxygen species (ROS), i.e. superoxide anion and hydroxyl radical. The potential therapeutic role of antioxidants in the chemoprevention of lung cancer has therefore been brought to major clinical trials in recent years. Disappointingly, the major landmark chemoprevention trials including the Alpha-Tocopherol, Beta Carotene Cancer Prevention (ATBC) study and the Beta-Carotene and Retinol Efficacy Trial (CARET) have failed to demonstrate therapeutic benefits of vitamins A and E in lung cancer. Apart from the criticism about the dosages being used in the trials, these results may reflect the lack of understanding of the exact role of antioxidants in lung carcinogenesis. The simple use of general antioxidants, vitamins A and E, may not be able to target specifically the peculiar alterations in antioxidant profiles that lead to the development of lung cancer. In fact, our recent study has demonstrated specific changes in antioxidant expressions in surgically resected non-small cell lung cancer. In the resected lung cancer tissues, there were increased manganese superoxide dismutase (Mn SOD) and decreased catalase expressions at the transcriptional levels as compared with adjacent normal lung tissues. It has been hypothesized that this alteration in local antioxidant levels may result in anti-apoptosis and accumulation of genetic damages thus perpetuating carcinogenesis. However the exact clinical implications are still under investigation. Our previous case-control study on the systemic (erythrocyte) antioxidant activities in patients with NSCLC has shown an increased glutathione peroxidase (GPx), but decreased SOD activities compared with healthy controls. The erythrocyte SOD activity was associated with disease staging. In addition, our recent study on longitudinal profile of erythrocyte antioxidants during chemotherapy for advanced NSCLC has identified total glutathione as an independent predictor to treatment response, which may reflect tumour load (submitted, unpublished data).

Exhaled breath condensate (EBC) has recently emerged as a non-invasive sampling method for real-time analysis and evaluation of oxidative stress biomarkers in the lower respiratory tract airways, especially in various lung diseases including asthma, chronic obstructive pulmonary disease, and lung cancer. In particular, endothelin-1 and interleukin-6 have been found to be elevated in the EBC from patients with lung cancer. Therefore, the current study aims to evaluate the temporal changes of various oxidative stress biomarkers and cytokines in EBC and blood in patients with NSCLC who are undergoing surgical lung resections and the potential role of these parameters in predicting subsequent tumour recurrence. Also, the correlation of biomarkers in blood or EBC with lung tumour tissue will be looked into.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed early-stage non-small cell lung cancer undergoing curative surgical lung resections.
* Life expectancy > 12 weeks.

Exclusion Criteria:

* Respiratory failure requiring use of supplemental oxygen therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early stage NSCLC who undergo curative lung resections in the Division of Cardiothoracic Surgery, Department of Surgery, Queen Mary Hospital will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2008-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to disease recurrence | 24 months after surgery

SECONDARY OUTCOMES:
Disease-free survival | 24 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chung-man James Ho, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong